CLINICAL TRIAL: NCT00179374
Title: Improving Diabetes Medication Adherence and Outcomes
Brief Title: Improving Diabetes Outcomes With Activity, Nutrition and Medication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Elizabeth Walker, Prof., Dept of Medicine, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2003-068; R18DK062038 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Medication adherence; Self-care behaviors; Telephonic intervention; Diabetes; Nutrition; Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tailored telephone intervention plus mailed print educational materials
  Interventions: Behavioral: Tailored telephone intervention of education
- 2 (Active Comparator): print intervention with no telephone component
  Interventions: Behavioral: Print educational intervention

INTERVENTIONS:
Behavioral: Tailored telephone intervention of education — Tailored telephone intervention to promote metabolic control of diabetes
  Arms: 1
Behavioral: Print educational intervention — diabetes educational materials by mail
  Arms: 2

SUMMARY:
This study has the following specific aims:

1. A tailored telephone intervention will significantly improve medication adherence compared to a standard care intervention.
2. A tailored telephone intervention will significantly improve metabolic control measured by HbA1c compared to a standard care intervention 2a) We will explore ways to link behavior change for medication adherence with lifestyle modification for diet and physical activity.
3. To conduct cost evaluations for the telephone intervention vs. standard care.

DETAILED DESCRIPTION:
Metabolic control of type 2 diabetes and prevention of its complications are related to management of blood glucose and other factors. Medication and lifestyle modifications are integral to most self-management plans; however, adherence remains a great challenge. Many patients have abnormal HbA1c, blood pressure and lipid values, and are at greater risk for complications. This study is to evaluate the effectiveness and costs of a tailored, telephone intervention to promote adherence in middle-aged and older adults with type-2 diabetes who are members of a union/employer-sponsored health benefit plan. The target population includes English- and Spanish-speaking individuals from the health plan database.

This study has the following specific aims:

1. A tailored telephone intervention will significantly improve medication adherence compared to a standard care intervention.
2. A tailored telephone intervention will significantly improve metabolic control measured by HbA1c compared to a standard care intervention 2a) We will explore ways to link behavior change for medication adherence with lifestyle modification for diet and physical activity.
3. To conduct cost evaluations for the telephone intervention vs. standard care. The study design is a randomized, controlled intervention trial with masking; the individual is the unit of sampling, assignment and analysis. After eligibility is assessed and consent is obtained by telephone, patients will be randomized to either the telephone intervention or standard are. Study outcomes will be medication adherence as measured from pharmacy records and metabolic control (HbA1c). A total of 556 patients with type 2 diabetes wil be randomized, which will provide 80% power to detect a statistically significant difference in HbA1c of at least 0.3%, and over 95% power to detect a difference in filled prescriptions. Telephone surveys will provide data on self-care behaviors including diet and exercise, risk perceptions, and depressive symptoms. Cost data will be collected using standardized methods. Study results will inform implementation of practical, nurse-managed interventions to improve medication adherence and metabolic control in diverse, middle-aged and older, type 2 diabetes patients, while linking changes in medication adherence to lifestyle modification for diet and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Taking oral diabetes medication
* At least 40 years old
* In a union-sponsored health plan with full medication coverage for at least a year
* Able to understand English or Spanish
* Informed consent

Exclusion Criteria:

* Currently in a diabetes education program
* Will lose health care eligibility within a year
* Unable to receive phone calls or mail

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2003-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 1 year
Metabolic control (measured by HbA1c) | 1 year

SECONDARY OUTCOMES:
Changes in self-care behaviors including diet and exercise | 1 year
Cost evaluations | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Walker, DNSc, RN, Principal Investigator — Albert Einstein College of Medicine; Hillel W Cohen, DrPH, MPH, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States